CLINICAL TRIAL: NCT04777916
Title: A Prospective Non-interventional Study Documenting the Management and Outcomes of Adult Patients With Acute Myeloid Leukemia (AML)
Brief Title: Prospective Non-interventional Study of Adult Patients With Acute Myeloid Leukemia (AML)
Acronym: ALFAPPP
Status: Recruiting | Type: Observational
Sponsor: Acute Leukemia French Association (Other)
Responsible Party: Sponsor
Other Study IDs: ALFA PPP Study
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Peripheral blood and bone marrow samples will be collected. Cells, and nucleic acids will be cryopreserved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Standard intensive 3+7 YOUNG OR ELDERLY: Standard intensive 3+7 (anthracycline + cytarabine) chemotherapy ± an approved FLT3 inhibitor (midostaurine, Rydapt® or ± quizartinib, Vanflyta®), according to different dose schedules in older versus younger patients
- GO, (Mylotarg®) with 3+7: Combination of sequential gemtuzumab ozogamicin (GO, Mylotarg®) with 3+7
- CPX-351, (Vyxeos®): Liposomal formulation of daunorubicin + cytarabine (CPX-351, Vyxeos®)
- Less intensive chemotherapy with azacytidine combined or not with venetoclax; LDAC; ivosidenib: Less intensive chemotherapy with azacytidine either combined or not with venetoclax or low dose cytarabine (LDAC) or in AML bearing an IDH1 somatic mutation, with ivosidenib in newly diagnosed patients considered as not eligible for the more intensive options above
- Refractory or relapsed AML: Secondly, no specific salvage regimen has emerged as a standard in patients with primary refractory or relapsed AML (R/R AML). R/R AML is thus an important field for investigational new drugs (INDs) and precision medicine development. To date, the only IND approved to treat R/R AML is gilteritinib for FLT3-mutated AML patients. The French agency ANSM also allow to use GO for treating R/R AML patients in the frame of a RTU (Recommendation Temporaire d'Utilisation).
  In the "real life", because of the multiplicity of treatments used in these patients, some of them being now quite efficient, it has become difficult to accurately describe the general outcome of R/R AML patients.

SUMMARY:
During the last fifteen years, the landscape of AML diagnosis and therapeutical options has markedly evolved. Refined genetic and prognostic characterizations, together with new drug approvals and new allogeneic hematopoietic stem cell transplantation (HSCT) procedures, have increased patient journey diversity.

DETAILED DESCRIPTION:
During the last fifteen years, the landscape of AML diagnosis and therapeutical options has markedly evolved. Refined genetic and prognostic characterizations, together with new drug approvals and new allogeneic hematopoietic stem cell transplantation (HSCT) procedures, have increased patient journey diversity.

I - At initial AML diagnosis, not all newly diagnosed patients are entering clinical trials. A substantial proportion of them are treated with standard therapies outside of any trial. To date, the standard approved frontline treatment options include:

1. Standard intensive 3+7 (anthracycline + cytarabine) chemotherapy ± an approved FLT3 inhibitor (midostaurine, Rydapt®), or ± quizartinib (Vanflyta®) according to different dose schedules in older versus younger patients
2. Combination of sequential gemtuzumab ozogamicin (GO, Mylotarg®) with 3+7
3. Liposomal formulation of daunorubicin + cytarabine (CPX-351, Vyxeos®)
4. Less intensive chemotherapy with azacytidine or low dose cytarabine (LDAC) in patients considered as not eligible for the more intensive options above

The investigator's choice is guided by AML and patient's characteristics, and by the approved indications for each of these treatment options. This study will thus start including these specific options. Further study amendments might be necessary in case of new standard treatment definition.

II - Secondly, no specific salvage regimen has emerged as a standard in patients with primary refractory or relapsed AML (R/R AML). R/R AML is thus an important field for investigational new drugs (INDs) and precision medicine development. To date, the only IND approved to treat R/R AML is gilteritinib for FLT3-mutated AML patients. The French agency ANSM also allow to use GO for treating R/R AML patients in the frame of a RTU (Recommendation Temporaire d'Utilisation).

In the "real life", because of the multiplicity of treatments used in these patients, some of them being now quite efficient, it has become difficult to accurately describe the general outcome of R/R AML patients.

III - Thirdly, allogeneic HSCT is no more considered at the ultimate and final goal of AML therapy in all patients, as it was in the past. Transplant indications have been better described and HSCT in now evaluated in the context of the whole treatment course, including pre- and post-transplant therapy, as well as pre- and post-transplant minimal residual disease (MRD) levels.

For all these reasons, it is of utmost importance to document the various characteristics, treatments and outcomes of patients treated in the real-life, outside of clinical trials, for 1) real-world treatment evaluation; 2) post-approval use of recently approved drugs; 3) standardization and improvement of routine patient management; and 4) better disease understanding.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years old or more
* Patient with newly diagnosed previously untreated de novo, secondary or therapy-related AML
* Patients with R/R de novo, secondary or therapy-related AML
* Patient with Health insurance

Exclusion Criteria:

* Acute promyelocytic leukemia
* AML which is not morphologically proven (patients with granulocytic sarcoma may be included)
* For newly diagnosed AML: previous treatment of leukemia apart from hydroxyurea. Previous anti leukemia treatments are allowed if they were administered before the diagnosis of AML to treat a MDS, MPN, MPN/MDS or CML
* Patient weighting less than 50 kgs
* Opposition of the patient to participate to this non-interventional study

More specific eligibility criteria might be requested to enter some study modules

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Natural History and assessment of the outcomes of different standard approved treatments in recently diagnosed or relapsed/refractory AML patients
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2032-04-01 (Estimated); Study Completion 2046-04-01 (Estimated)

PRIMARY OUTCOMES:
OS | 1 year
  The primary objective of this multicenter non-interventional study is to record and prospectively evaluate the real-life characteristics, treatments and outcomes of adult patients with newly diagnosed or R/R AML, when managed and treated in the French ALFA centers according to standard practices outside of a clinical trial.
  The two co-primary endpoints are event-free (EFS) and overall survival (OS) estimations at 1, 3, 5 and 10 years:
  * From first treatment initiation in patients with newly diagnosed AML
  * From the date of relapse/refractoriness (R/R) in patients, with R/R AML
OS | 3 years
  The primary objective of this multicenter non-interventional study is to record and prospectively evaluate the real-life characteristics, treatments and outcomes of adult patients with newly diagnosed or R/R AML, when managed and treated in the French ALFA centers according to standard practices outside of a clinical trial.
  The two co-primary endpoints are event-free (EFS) and overall survival (OS) estimations at 1, 3, 5 and 10 years:
  * From first treatment initiation in patients with newly diagnosed AML
  * From the date of relapse/refractoriness (R/R) in patients, with R/R AML
OS | 5 years
  The primary objective of this multicenter non-interventional study is to record and prospectively evaluate the real-life characteristics, treatments and outcomes of adult patients with newly diagnosed or R/R AML, when managed and treated in the French ALFA centers according to standard practices outside of a clinical trial.
  The two co-primary endpoints are event-free (EFS) and overall survival (OS) estimations at 1, 3, 5 and 10 years:
  * From first treatment initiation in patients with newly diagnosed AML
  * From the date of relapse/refractoriness (R/R) in patients, with R/R AML
OS | 10 years
  The primary objective of this multicenter non-interventional study is to record and prospectively evaluate the real-life characteristics, treatments and outcomes of adult patients with newly diagnosed or R/R AML, when managed and treated in the French ALFA centers according to standard practices outside of a clinical trial.
  The two co-primary endpoints are event-free (EFS) and overall survival (OS) estimations at 1, 3, 5 and 10 years:
  * From first treatment initiation in patients with newly diagnosed AML
  * From the date of relapse/refractoriness (R/R) in patients, with R/R AML
EFS | 1 year
  The primary objective of this multicenter non-interventional study is to record and prospectively evaluate the real-life characteristics, treatments and outcomes of adult patients with newly diagnosed or R/R AML, when managed and treated in the French ALFA centers according to standard practices outside of a clinical trial.
  The two co-primary endpoints are event-free (EFS) and overall survival (OS) estimations at 1, 3, 5 and 10 years:
  * From first treatment initiation in patients with newly diagnosed AML
  * From the date of relapse/refractoriness (R/R) in patients, with R/R AML
EFS | 3 years
  The primary objective of this multicenter non-interventional study is to record and prospectively evaluate the real-life characteristics, treatments and outcomes of adult patients with newly diagnosed or R/R AML, when managed and treated in the French ALFA centers according to standard practices outside of a clinical trial.
  The two co-primary endpoints are event-free (EFS) and overall survival (OS) estimations at 1, 3, 5 and 10 years:
  * From first treatment initiation in patients with newly diagnosed AML
  * From the date of relapse/refractoriness (R/R) in patients, with R/R AML
EFS | 5 years
  The primary objective of this multicenter non-interventional study is to record and prospectively evaluate the real-life characteristics, treatments and outcomes of adult patients with newly diagnosed or R/R AML, when managed and treated in the French ALFA centers according to standard practices outside of a clinical trial.
  The two co-primary endpoints are event-free (EFS) and overall survival (OS) estimations at 1, 3, 5 and 10 years:
  * From first treatment initiation in patients with newly diagnosed AML
  * From the date of relapse/refractoriness (R/R) in patients, with R/R AML
EFS | 10 years
  The primary objective of this multicenter non-interventional study is to record and prospectively evaluate the real-life characteristics, treatments and outcomes of adult patients with newly diagnosed or R/R AML, when managed and treated in the French ALFA centers according to standard practices outside of a clinical trial.
  The two co-primary endpoints are event-free (EFS) and overall survival (OS) estimations at 1, 3, 5 and 10 years:
  * From first treatment initiation in patients with newly diagnosed AML
  * From the date of relapse/refractoriness (R/R) in patients, with R/R AML

CONTACTS AND LOCATIONS:
Overall Officials: Hervé DOMBRET, PD-Prof, Study Chair — Acute Leukemia French Association
Locations (30):
- France (30):
  - Chu Amiens, Amiens
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - AP-HP-GHU - Hôpital AVICENNE, Bobigny
  - CHU de la cote de Nacre, Caen
  - Hôpital MILITAIRE PERCY, Clamart
  - Centre hospitalier Sud Francilien, Corbeil-Essonnes
  - Hôpital Henri Mondor AP-HP, Créteil
  - CHU Dijon- François Mitterrand, Dijon
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Centre Hospitalier de Versailles André Mignot, Le Chesnay
  - Centre Hospitalier Dr Schaffner, Lens
  - CHRU de Lille- Hopital C. HURIEZ, Lille
  - GHICL-Hopital St Vincent de Paul, Lille
  - C H U DE LIMOGES- Hopital Dupuytren, Limoges
  - CHU La Conception, Marseille
  - Centre Hopsitalier de l'Est Francilien - Site de Meaux, Meaux
  - Centre Antoine Lacassagne, Nice
  - CHU Nice,Hopital Archet 1, Nice
  - Hopital Pitié-Salpétrière APHP, Paris
  - Hôpital Necker - APHP, Paris
  - Hôpital SAINT ANTOINE-APHP, Paris
  - Hôpital Saint Louis- APHP, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier René Dubos, Pontoise
  - Centre Hospitalier de Roubaix, Roubaix
  - Centre Henri Becquerel, Rouen
  - Institut Curie - Hôpital René HUGUENIN, Saint-Cloud
  - Centre Hospitalier de St Quentin, Saint-Quentin
  - Centre Hospitalier Valenciennes, Valenciennes
  - Institut Gustave Roussy, Villejuif